CLINICAL TRIAL: NCT03531034
Title: Ambulatory and Blood Pressure Variability Responses to Combined Exercise in Normotensive and Hypertensive Menopausal Women
Brief Title: Ambulatory and Blood Pressure Variability Responses to Exercise in Normotensive and Hypertensive Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Uberlandia (Other)
Responsible Party: Principal Investigator, Igor Moraes Mariano, Principal Investigator, Federal University of Uberlandia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 40622414.9.0000.5152
Record Dates: First submitted 2018-04-17; First posted 2018-05-21 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Menopause; Exercise; Blood Pressure, High
Keywords: Blood Pressure Variability; Ambulatorial Blood Pressure Monitoring; Combined Exercise
MeSH Terms: conditions — Motor Activity; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertensive Women (Experimental): Group of hypertensive and controlled women who practiced 10 weeks of training with Combined Exercise Training, non-obese, nonsmokers and with no characteristics that prevented them from performing the activities. In addition this group could not modify the dose or type of the medicine and should be using the same medicine and dose for at least 6 months
  Interventions: Other: Combined Exercise Training
- Normotensive Women (Active Comparator): Group of normotensive women who practiced 10 weeks of training with Combined Exercise Training, non-obese, nonsmokers and with no characteristics that prevented them from performing the activities.
  Interventions: Other: Combined Exercise Training

INTERVENTIONS:
Other: Combined Exercise Training — The program consisted of 30 sessions of combined aerobic and resistance exercises training during 10 consecutive weeks. Each session lasted 45 minutes and consisted of 5 minutes warm-up, 20 minutes of resistance exercise and 20 minutes of aerobic exercise. The resistance training was performed in two sets of 15 repetitions in seven exercises of weight training (Based on 1 repetition maximum test - 1RM) for large muscle groups. The aerobic exercise was performed on a treadmill, at a speed of 5.5 km/h and intensity (imposed by treadmill inclination and heart rate) between ventilatory threshold 1 and 2 intensities. After 5 weeks of training, 1RM test was performed again to readjust the resistance load and aerobic intensity was readjusted by heart rate predicted in the incremental test.

SUMMARY:
This study evaluated the differences between normotensive and hypertensive menopausal women in ambulatory and blood pressure variability responses to combined aerobic and resistance exercise.

DETAILED DESCRIPTION:
The differences in hypotensive and cardioprotective responses of exercise among menopausal hypertensive and normotensive women are still not very clear, mainly the responses of blood pressure variability. In this way, were evaluated 6 indices related to the variability of 24 hour ambulatory pressure measurements in these women before and after 12 weeks of combined exercise training.

ELIGIBILITY:
Inclusion Criteria:

* amenorrhea for at least 12 months; body mass index ≤30 kg/m2; ability to engage in treadmill and resistance exercises; hypertension nom-medicated with beta-blockers

Exclusion Criteria:

* history of diabetes, cancer or cardiovascular disease (except for hypertension in Hypertensive group); doing hormone therapy or soy derived supplementation; smokers

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2015-12-25 (Actual); Study Completion 2016-12-25 (Actual)

PRIMARY OUTCOMES:
Changes in Ambulatorial Blood Pressure | Before and within 72 hours after 10 weeks of exercise training
  All volunteers were submitted to a 24-hour Blood Pressure (BP) assessment by Ambulatorial Blood Pressure Monitoring (ABPM) before and after 10 weeks of combined exercise training, with a minimum of 48 hours after the last training session. A device was used associated with a diary of examination to self-report of activities of daily living (sleep, work, food) or any event that could interfere abnormally with BP or device measurements. The device was always placed 7am and the measurements were made every 15 minutes from 7h to 23h and every 30 minutes from 23h to 7h. The monitoring was considered valid when it happened for a period of 24 hours. The following results were evaluated: systolic blood pressure; diastolic blood pressure, mean blood pressure and heart rate in awake, sleep and 24-hour periods. Before the use ABPM during daily activities, resting blood pressure were measured using the same equipment after 15 min of rest in siting position.

SECONDARY OUTCOMES:
Changes in Ambulatorial Blood Pressure Variability | Before and within 72 hours after 10 weeks of exercise training
  Based on Ambulatorial Blood Pressure data, were calculated Blood Pressure Variability by: 24-hour standard deviation weighted by the time interval between consecutive readings; the mean diurnal and nocturnal deviations weighted for the duration of the daytime and nighttime interval; the average real variability weighted for the time interval between consecutive readings; the ambulatory arterial stiffness index calculated by the slope of the trend curve of the dispersion of pressure data; the morning surge that represents the dynamic daytime variation in morning pressure that tends to increase, being assessed from the point of least pressure during sleep in relation to the first two hours after waking; and nocturnal dipping, that represents the average percentage drop of sleep pressure in relation to wakefulness, and individuals with falls of 10% or more are considered dippers and below that are considered nom-dippers.
Changes in Heart Rate Variability | Before and within 72 hours after 10 weeks of exercise training
  Heart Rate (HR) was recorded using a heart rate monitor in a beat-by-beat basis. HR was registered in a seat position for 20 min of rest. Prior to the HR Variability (HRV) analysis, the RR intervals (RRi) were visually inspected and filtered using a moving average filter. The HRV was analyzed in both time-, frequency- and nonlinear-domain. Being that for frequency-domain analysis, firstly the RRi series were interpolated at 4 Hz and then the signal linear trend component removal was performed using the smooth priors approach.
Changes in salivary oxidative stress | Before and within 72 hours after 10 weeks of exercise training
  The salivary was collected after 12-hours fasting and the total antioxidant capacity was evaluated using the Ferric-Ability of Plasma (FRAP) methodology and calculated from the standard trolox curve. The activity of the enzyme superoxide dismutase (SOD) was determined based on the auto oxidation capacity of pyrogallol and catalase activity (CAT) by monitoring the consumption of hydrogen peroxide at 240 nm. Lipid peroxidation levels were determined by the TBARS method (thiobarbituric acid reactive substances), using as standard a curve of 1,1,3,3-tetraethoxypropane (TMP). The total protein concentration was obtained by the Bradford method (BRADFORD, 1976), using bovine serum albumin (BSA) as standard. The amounts of nitric oxide (NO) were estimated by the determination of total nitrite by the Griess colorimetric method.

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme M Puga, Dr, Principal Investigator — Federal University of Uberlandia
Locations (1):
- Guilherme Morais Puga, Uberlândia, Minas Gerais, Brazil